CLINICAL TRIAL: NCT02187913
Title: Effects of Resistant Starch in a Baked Snack Bar on a Post-prandial Glycemic and Insulinemic Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1406014929
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Hyperglycemia, Diabetes, and Obesity
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus; Obesity | interventions — Resistant Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resistant starch (Experimental): The test snack bar consumed has the resistant starch
  Interventions: Dietary Supplement: Resistant starch
- Control (Experimental): The control bar uses maltodextrin rather than the resistant starch.
  Interventions: Dietary Supplement: Resistant starch

INTERVENTIONS:
Dietary Supplement: Resistant starch — Each subject will complete 2 testing days (randomized and crossover design). On each of 2 test days, subjects will arrive at the Purdue Clinical Research Center after a 12-h fast and will consume a snack bar containing resistant starch. The test snack bar will be consumed along with a standard meal provided at the start of the test day. A second standard meal that does not contain the snack bar will be consumed four hours later.

SUMMARY:
* About two-thirds of adults in the United States are overweight or obese which can cause adverse health consequences for those individuals. Post-prandial hyperglycemia is one of these possible consequences and is associated with a higher risk for Type 2 Diabetes. Controlling hyperglycemia is important in the prevention of the onset of diabetes and obesity. Resistant starch is a dietary carbohydrate which is not completely digested in the gut and produces energy for the body to use. The investigators are interested in assessing the effects of resistant starch on postprandial blood glucose and insulin concentrations.
* Aim: To assess the effects of a resistant starch on post-prandial blood glucose and insulin concentrations.
* Hypothesis: A baked snack bar with a resistant starch will blunt and sustain the post-prandial rise in blood glucose and insulin concentrations compared to a baked snack bar with maltodextrin (an easily digested carbohydrate).

ELIGIBILITY:
Inclusion Criteria:

* Thirty healthy men and women (aged 18-29y) will be recruited from the greater Lafayette, IN region with the expectation that ≥20 subjects will complete the study. Subjects must weigh >110 pounds, with a BMI between 20.0 and 29.9.

Exclusion Criteria:

* Weight change > 3kg in the past 3 months
* Exercising vigorously over the past 3 months as well as no exercise 3 days prior to testing day
* Intestinal disorders including lipid mal-absorption or lactose intolerance
* Abnormal liver or kidney function tests; fasting blood glucose >100mg/dL
* Smoking
* Drinking more than 2 alcoholic drinks per day
* Taking lipid-lowering medications or dietary supplements affecting plasma cholesterol concentration.
* Subjects must not be pregnant or lactating.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
resistant starch effects | 2 weeks
  effects of resistant starch consumption of area under the curve of blood serum glucose, insulin, and hydrogen breath testing

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States